CLINICAL TRIAL: NCT04968106
Title: Randomized Phase II Study of Neoadjuvant Chemotherapy Plus Retifanlimab (INCMGA00012) in Patients With Selected Sarcomas
Brief Title: Neoadjuvant Chemotherapy and Retifanlimab in Patients With Selected Sarcomas (TORNADO)
Acronym: TORNADO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2021-01; 2021-001085-37 (EudraCT Number)
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Resectable Sarcoma
Keywords: sarcoma; neoadjuvant chemotherapy; mature tertiary lymphoid structures; immune checkpoint inhibitor
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, open-labeled, 2-arm, non-comparative randomized (1:1) phase II trial. Patients will be randomized between arm A (neodjuvant chemotherapy by doxorubicin + ifosfamide) and arm B (neodjuvant chemotherapy by doxorubicin + ifosfamide and retifanlimab) with one patient randomized in arm A for one patient randomized in arm B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm A: treatment by neoadjuvant chemotherapy (Other): Treatment by doxorubicin and ifosfamide followed by surgery
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide
- Experimental Arm B: treatement by neoadjuvant chemotherapy and retifanlimab (Experimental): Treatment by doxorubicin, ifosfamide and retifanlimab followed by surgery
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide; Drug: INCMGA00012

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin will administered by intravenous infusion on day 1 every 3 weeks (75 mg/m²) up to 3 cycles
Drug: Ifosfamide — Ifosfamide will be administered by intravenous infusion over 3 days every 3 weeks (9 g/m²) up to 3 cycles
Drug: INCMGA00012 — Retifanlimab will be administered by intravenous infusion on day 1every 3 weeks (375 mg) up to 3 cycles
  Other Names: Retifanlimab
  Arms: Experimental Arm B: treatement by neoadjuvant chemotherapy and retifanlimab

SUMMARY:
Multicenter, prospective, open-labeled, 2-arm, non-comparative randomized phase II trial to assess the antitumor activity of retifanlimab (INCMGA00012) in association with neoadjuvant chemotherapy

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-labeled, 2-arm, non-comparative randomized (1:1) phase II trial. Patients will be randomized between arm A (neodjuvant chemotherapy by doxorubicin + ifosfamide) and arm B (neodjuvant chemotherapy by doxorubicin + ifosfamide and retifanlimab) with one patient randomized in arm A for one patient randomized in arm B.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with grade 2 or grade 3 soft-tissue sarcoma (limb, trunk wall, retroperitoneum) histologically confirmed and reviewed by the RRePS Network
2. For TLS status determination: available archived FFPE tumor tissue sample.
3. Presence of mature tertiary lymphoid structures. Except if presence of TLS have been already confirmed by Biopathological platform at Bergonié Institute, presence of TLS should be confirmed by central review based on FFPE tumor tissue sample (archived or newly obtained by biopsy for research purpose).
4. Non-metastatic and resectable disease,
5. At least one lesion that can be biopsied for research purpose,
6. No prior treatment for the disease under study,
7. Age ≥ 18 years,
8. ECOG ≤ 1,
9. Life expectancy > 3 months,
10. Patients must have measurable disease defined as per RECIST v1.1
11. Adequate hematological, renal, metabolic and hepatic function
12. Left ventricular ejection fraction ≥ 50% assessed by ECHO or MUGA within 6 months from study entry,
13. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to study entry. .
14. Both women and men must agree to use a highly effective method of contraception throughout the treatment period and for one year after discontinuation of treatment for women and 4 months for men.
15. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, concomitant endometrial carcinoma stage IA grade 1, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
16. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5),
17. Voluntarily signed and dated written informed consent prior to any study specific procedure,
18. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Previous treatment for retroperitoneal sarcoma including surgery, chemotherapy or radiotherapy
2. Previous treatments with doxorubicin, daunorubicin, epirubicin, idarubicin and/or other anthracyclines or anthracenediones at the maximum cumulative dose,
3. Known hypersensitivity to any involved study drug or any of its formulation components,
4. Has an active or ongoing infection requiring systemic therapy,
5. Known central nervous system malignancy (CNS),
6. Women who are pregnant or breast feeding,
7. Has known active hepatitis B or hepatitis C,
8. Has a known history of Human Immunodeficiency Virus (HIV),
9. Previous enrolment in the present study,
10. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
11. Has received a live attenuated vaccine or a live vaccine within 30 days prior to the first dose of trial treatment, Note: the killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
12. Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

    1. Myocardial infarction or stroke/transient ischemic attack within the 6 months prior to study entry.
    2. Uncontrolled angina within the 3 months prior to study entry.
    3. Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes, or poorly controlled atrial fibrillation).
    4. Corrected QT (QTc) prolongation > 480 msec.
    5. History of other clinically significant cardiovascular disease (i.e., cardiomyopathy, congestive heart failure with New York Heart Association [NYHA] functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled venous thrombus).
13. Uncontrolled or significant renal disease including, but not limited to, any of the following:

    1. Acute or uncontrolled urinary infection at study entry,
    2. Hemorrhagic cystitis at study entry,
    3. Presence of blood on dipstick at study entry,
    4. Vesical atony,
    5. Known urinary tract obstruction.
14. Patients with known history of active inflammatory bowel diseases, including those with small or large intestine inflammation, such as Crohn's disease or ulcerative colitis, will be excluded from the study,
15. Has received systemic antibiotics within 14 days before the first dose of study treatment. Participants receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
16. History of organ transplant, including allogeneic stem cell transplantation.
17. Receiving probiotics as of the first dose of study treatment.
18. Has an active autoimmune disease

    * Patients with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible,
    * Patients requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at dose ≤ 10 mg or 10 mg equivalent prednisone day,
    * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intra-ocular, intra-articular or inhalation) are acceptable.
19. Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis.
20. Palliative radiation therapy administered within 1 week of first dose of study treatment or radiation therapy in the thoracic region that is > 30 Gy within 6 months of the first dose of study treatment. Note: Participants must have recovered from all radiation-related toxicities (to Grade >1 or baseline), not require corticosteroids for this purpose, and not have had radiation pneumonitis.
21. Person under judicial protection or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of retifanlimab when prescribed in association with neoadjuvant chemotherapy (doxorubicin+ifosfamide) | 5 months after treatment onset
  Antitumor activity will be assessed in terms of histological response based on surgical sample

SECONDARY OUTCOMES:
1-year progression-free survival | 1 year
  Progression-free survival (PFS) is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
3-year progression-free survival | 3 years
  Progression-free survival (PFS) is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
1-year overall survival | 1 year
  Overall Survival (OS) is defined as the time from study treatment initiation to death (of any cause).
3-year overall survival | 3 years
  Overall Survival (OS) is defined as the time from study treatment initiation to death (of any cause).
Safety profile independently for each arm: Common Terminology Criteria for Adverse event version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity will be grade using the Common Terminology Criteria for adverse events version 5 and coded according to the standardized medical terminology MedDRA

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No